CLINICAL TRIAL: NCT00729781
Title: Open Label, Baseline Controlled Study to Evaluate the Use of Polyethylene Terephthalate (PET) Implants for the Treatment of External Nasal Valve Collapse and Cosmetic Contour Deformity
Brief Title: Study of Polyester Implants for the Treatment of External Nasal Valve Collapse (NVC)
Acronym: NVC
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Medtronic Xomed, Inc. (Industry)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 925
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2012-01-06 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2011-12

CONDITIONS: Nasal Alar Collapse, Bilateral
Keywords: nasal obstruction; airway resistance; soft tissue collapse; cosmetic contour deformity
MeSH Terms: conditions — Nasal Alar Collapse, Bilateral; Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Polyester Implants (Experimental): There is one arm for this study. All subjects in this study will receive the investigational nasal implants. See the detailed description for procedure information.
  Interventions: Device: Polyester Implants

INTERVENTIONS:
Device: Polyester Implants — Three polyester (PET) implants will be implanted in each side of the nose affected by external NVC. See the detailed description for information about the implant procedure.
  Other Names: NVC-1000; The Pillar(R) Procedure; Pillar(R) Palatal Implants

SUMMARY:
The purpose of this study is to research a polyester polyethylene terephthalate (PET) implant for the treatment of external nasal valve collapse (NVC). NVC is a condition which causes narrowness and weakness in the nostril which results in nasal obstruction. Implants will be placed in the affected nostril(s). The implants are intended to restore the shape and stabilize the nasal wall to prevent nasal valve collapse and improve the symptoms associated with nasal obstruction.

DETAILED DESCRIPTION:
The effects of PET implants on external NVC and cosmetic contour deformity will be evaluated in an open-label, prospective study. Subjects for this clinical study will be recruited and screened from clinic office visits and patient records at each principal investigator's site as well as through an investigational review board (IRB)-approved general advertisement. Those patients that continue to qualify after either screening process will be seen and evaluated by one of the clinical investigators prior to enrollment in the study. Subjects must meet criteria for the diagnosis of external nasal valve collapse as a stand alone abnormality (i.e., symptoms of obstruction cannot be caused primarily by other factors). Other contributing factors to the nasal obstruction must be ruled out and/or treated, without relief before enrollment in this study. No other surgeries or procedures will be allowed during the study that could influence the evaluation of implants on the treatment of nasal valve collapse and cosmetic contour deformity. All subjects will be required to sign an IRB approved informed consent prior to entry into the study.

After meeting inclusion/exclusion criteria and completing the pre-implant evaluations, subjects will be scheduled for treatment with the polyethylene terephthalate implants. The implant procedure will be performed by facial plastic physicians. All investigative sites will be required to undergo training to standardize the methodology of implant technique and administration of evaluation techniques (questionnaires, scales, photographic assessments, etc.). Target sample size for the study will be 72 subjects.

Follow up evaluations for all outcome measures will occur at 1, 6, and 12 weeks after implantation. Long-term follow-up for adverse events will be conducted at 11 months or later after implantation.

ELIGIBILITY:
Inclusion Criteria:

* Is willing and able to sign an informed consent form
* Is 18 years of age or older
* Has positive response to any of the following based on patient history or office exam:

  * Use of Breath Rite Strips
  * Q-Tip test
  * Use of Nasal stents
  * Continuous manual distraction
* Has inspiratory lateral nasal wall collapse or static medially obstructing lateral nasal wall position identified on physical exam
* Has nasal valve that is narrow (either static or dynamic) based on a visual examination.
* Has nasal septum that is considered stable and adequate to support the treatment of each nasal valve independently.
* Is motivated and willing to comply with study and its follow-up requirements, including surgical intervention using the Pillar implant system for the treatment of nasal valve collapse
* Speaks English
* Has unilateral or bilateral nasal valve collapse

Exclusion Criteria:

* Has ability to achieve active nostril dilation and relieve obstruction using physiologic nasal alar and sidewall muscle actions
* Has chronic sinusitis, recurrent sinusitis, or allergies leading to nasal obstruction.
* Has active nasal infection
* Has skin inflammation in the nasal area
* Is a habitual chronic sniffer
* Has septal deviation, turbinate hypertrophy, polyps, or ptotic nose tip believed to be causing obstruction
* Has had previous rhinoplasty of external nasal frame
* Requires another surgery other than implants to correct an obstruction
* Has nasal anatomy that is inadequate to accommodate three 18 mm implants
* Is participating in a clinical study for another treatment for nasal valve collapse
* Is pregnant or desires to become pregnant during the duration of the study
* Has a history of drug abuse or alcoholism in the year before enrollment
* Has had previous surgery for external nasal valve collapse
* Has an American Society of Anesthesiologists (ASA) rating of III or IV
* Has any other condition believed to interfere with nasal assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-04; Primary Completion 2009-11 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Terry L Donat, MD, Principal Investigator — Institute of Aesthetic Surgery
Locations (5):
- United States (5):
  - UC Davis Medical Center, Sacramento, California
  - Premier Image Cosmetic & Laser, Atlanta, Georgia
  - DuPage Medical Group, Ltd, Downers Grove, Illinois
  - Ear, Nose, & Throat Physicians, Sterling Heights, Michigan
  - HealthPartners Specialty Clinic/Regions Hospital, Saint Paul, Minnesota

REFERENCES:
- [Background] Hurbis CG. An adjustable, butterfly-design, titanium-expanded polytetrafluoroethylene implant for nasal valve dysfunction: a pilot study. Arch Facial Plast Surg. 2006 Mar-Apr;8(2):98-104. doi: 10.1001/archfaci.8.2.98. PMID 16549736
- [Background] Stewart MG, Witsell DL, Smith TL, Weaver EM, Yueh B, Hannley MT. Development and validation of the Nasal Obstruction Symptom Evaluation (NOSE) scale. Otolaryngol Head Neck Surg. 2004 Feb;130(2):157-63. doi: 10.1016/j.otohns.2003.09.016. PMID 14990910

RESULTS

PARTICIPANT FLOW:
Groups:
- Polyester Implants: There was one arm for this study. All subjects in this study received the investigational polyethylene terephthalate (PET) implants after enrollment in the original study. Subjects who could be reached and consented were enrolled in the long-term follow-up study, which was initiated to collect adverse events. See the detailed description for procedure information.
Period: Original Study
Arm/Group | Polyester Implants
Started | 45
Completed | 45
Not Completed | 0
Period: Long-term Follow-up Study
Arm/Group | Polyester Implants
Started | 42 (Enrollment in the long-term follow-up required contact and a new Informed Consent.)
Completed | 42 (All subjects completed the original study, but 3 did not consent to enroll in the follow-up study.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Polyester Implants
Number analyzed (Participants) | 45
Age Continuous [Mean (Standard Deviation); unit: years]
  All subjects | 45.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22
Race/Ethnicity, Customized [Number; unit: participants]
  White | 43
  Hispanic | 2

OUTCOME MEASURES:

1. Primary Outcome: Functional Improvement
Description: Functional improvement was defined as a subject who achieves both 1) an improvement in the physical condition of the collapsed nasal valve as evidenced by an increase of >= 10% in the change in volume during inspiration as measured by Vectra 3D photography from baseline to 12 weeks post-procedure; and 2) a reduction of at least 30% in the symptoms of nasal obstruction as measured by the Nasal Obstruction Symptom Evaluation Scale (NOSE) scale (5 questions with 0-4 scale from "Not a problem" to "Severe problem," possible score 0-100 via raw score × 5) from baseline to 12 weeks post-procedure.
Time Frame: 12 weeks after implantation
Population: An implanted subject with missing data at 12 weeks of follow-up had the 6-week data carried forward to 12 weeks for analysis. If the 6-week data was unavailable, the subject's treatment was considered a failure.
Measure: Number; unit: participants
Arm/Group | Polyester Implants
Number analyzed (Participants) | 45
participants
  ≥ 30% reduction in NOSE score | 40
  ≥ 10% increase in volume deflection (Vectra 3D) | 30
  ≥ 30% NOSE reduction and ≥ 10% Vectra 3D increase | 26
Statistical Analysis 1: Comparison: Polyester Implants; This study had two independent primary endpoints (cosmetic and functional improvement). Therefore, the assumed type I error rate for each was 2.5% in order to maintain an overall 5% type I error rate. For each endpoint, the percent of subjects with improvement of the total number implanted was to be compared to a rate of 50% using a one-sided, binomial exact test. If the p-value was < 0.025, the objective would have been met; Test type: Superiority or Other; p = 0.19, One-sided, binomial exact test; Percent of subjects with improvement = 57.8, 97.5% CI 1-sided [lower limit 42.2]

2. Primary Outcome: Cosmetic Improvement
Description: An independent clinician will review Vectra 3D photographs of each subject at baseline and at 12 weeks post-procedure to assess physical appearance of the external nasal wall. The clinician will be asked to determine which photographs are pre-treatment and which are post-treatment in the correct order. The clinician will then rate the photograph chosen as post-treatment using the Global Aesthetic Improvement Scale (GAIS; relative scale from "Worse" to "Very much improved"). If the post-treatment photograph was not correctly identified, that procedure will receive a "worse" on the rating scale.
Time Frame: 12 weeks after implantation
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Polyester Implants
Number analyzed (Participants) | 45
participants
  Order of photos: Could not evaluate | 11
  GAIS: Worse (After correct order ID) | 4
  GAIS: No change (After correct order ID) | 15
  GAIS: Improved (After correct order ID) | 7
  GAIS: Much improved (After correct order ID) | 0
  GAIS: Very much improved (After correct order ID) | 0
  GAIS: Could not evaluate (After correct order ID) | 0
  GAIS: Worse (After incorrect order ID) | 8
Statistical Analysis 1: Comparison: Polyester Implants; Test type: Superiority or Other; p > 0.99, One-sided, binomial exact test; Percent of subjects with improvement = 15.6, 97.5% CI 1-sided [lower limit 0.05]

3. Primary Outcome: Safety
Description: Evaluate complications and adverse events. Events are presented descriptively with no statistical analysis.
Time Frame: During 12-week original study and at long-term follow-up of 11 months or longer
Population: All enrolled subjects' adverse events were collected.
Measure: Number; unit: events
Arm/Group | Polyester Implants
Number analyzed (Participants) | 45
events
  Temporary pain implant site | 39
  Partial extrusion | 17
  Foreign body sensation | 11
  Upper respiratory infection/viral cold | 8
  Cosmetic contour deformity | 7
  Swelling/edema | 7
  Minimal bleeding | 4
  Cellulitis | 3
  Fever | 2
  Redness of skin | 2
  Tenderness | 2
  Vestibulitis | 2
  Sinus infection | 2
  Vomiting | 2
  Full extrusion | 1
  Infection | 1
  Bronchitis | 1
  Ecchymosis right cheek | 1
  Halitosis dysgusia | 1
  Herniated disc | 1
  Intranasal irritation/crust | 1
  Mild bruising perinasal | 1
  Numbness to tip of nose | 1
  Post inflammatory neuralgia | 1
  Pustule w/ implant exposure | 1
  Surface irritation sensation | 1
  Scarring | 1

ADVERSE EVENTS:
Arm/Group | Polyester Implants
Serious Adverse Events (participants affected / at risk) | 0/45
Other Adverse Events (participants affected / at risk) | 36/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Polyester Implants (N=45)
Temporary pain implant site (Skin and subcutaneous tissue disorders) | 28 (39)
Partial extrusion (Surgical and medical procedures) | 9 (17)
Foreign body sensation (Skin and subcutaneous tissue disorders) | 11 (11)
Upper respiratory infection/viral cold (Respiratory, thoracic and mediastinal disorders) | 7 (8)
Cosmetic contour deformity (Surgical and medical procedures) | 6 (7)
Swelling/edema (Skin and subcutaneous tissue disorders) | 7 (7)
Minimal bleeding (Surgical and medical procedures) | 3 (4)
Cellulitis (Skin and subcutaneous tissue disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days